CLINICAL TRIAL: NCT05255614
Title: Comparative Study to Determine Proper Sequence of Simulation Training Pelvic Versus Virtual Reality Simulator
Brief Title: Pelvic vs Virtual Reality Simulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Abdalla, Clinical professor of Obstetrics and Gynecology, Cairo University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Pelvic trainer vs VRS
Record Dates: First submitted 2022-01-19; First posted 2022-02-24 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Laparoscopic Training
Keywords: Simulation training; Pelvic trainer; Virtual reality Simulator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Group (Active Comparator): the participants will start training on the pelvic trainer and assessment will be via assessment via a checklist. Then at a later time, they will be trained on VR simulator (Sim Surgery) and assessment will be via Electronic auto assessment via the Simulator.
  Interventions: Device: Virtual reality Simulator; Device: Pelvic trainer:
- Second Group (Active Comparator): the participants will start training on VR simulator (Sim Surgery) and assessment will be via Electronic auto assessment via the Simulator. Then at a later time, they will be trained on the pelvic trainer and assessment will be via assessment via a checklist.
  Interventions: Device: Virtual reality Simulator; Device: Pelvic trainer:

INTERVENTIONS:
Device: Virtual reality Simulator — LapSim is a device designed by Surgical Science Device & software at Swedan
  Other Names: LapSim
Device: Pelvic trainer: — Video-box trainers include a box with a lid and holes cut on the lid for the trocar's insertion. A laparoscope inside the box is connected with a digital camera and provides video output to a monitor on which the trainees are watching their own movements, while performing the teaching task. Laparoscopic instruments, such as laparoscopic graspers and laparoscopic scissors are inserted through the trocars into the box, where the tasks are taught

SUMMARY:
The aim of this study is to evaluate the proper sequence of Pelvic trainer and VR simulator training in order to improve gynecological laparoscopic skills and assess training levels.

DETAILED DESCRIPTION:
In this study, the investigators will determine the proper sequence of simulation training. Pelvic Trainer Versus Virtual reality Simulator in order to improve laparoscopic skills of residents with no or little previous laparoscopic experience.

* This study will compare the proper sequence of simulation training. Pelvic Trainer Versus Virtual reality Simulator of two groups: Group A versus Group B.
* Group A will start training on the pelvic trainer (training on educational intervention 1) and assessment will be via assessment via a checklist (test 1). Then at a later time, they will be trained on VR simulator (Sim Surgery) (educational intervention 2) and assessment will be via Electronic auto assessment via the Simulator (test 2).
* Group B will start training on the VR simulator (Sim Surgery) (educational intervention 2) and assessment will be via Electronic auto assessment via the Simulator (test 2). Then at a later time, they will be trained on the pelvic trainer (training on educational intervention 1) and assessment will be via assessment via a checklist (test 1).

ELIGIBILITY:
Inclusion Criteria:

* All the residents in Obstetrics and Gynecology department who have no or little previous laparoscopic experience

Exclusion Criteria:

* Residents who have previous good laparoscopic experiences.
* Age below 26 or Above 29 years

Ages: 26 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
assessment of time needed to accomplish the tests before and after pelvic trainer | 6 months
  assessment of time needed to accomplish the tests before and after pelvic trainer
assessment of time needed to accomplish the tests before and after victual reality simulator | 6 months
  assessment of time needed to accomplish the tests before and after victual reality simulator

CONTACTS AND LOCATIONS:
Overall Officials: Marwa M Abdalla, MD, Principal Investigator — Kasralainy teaching hospital
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- See also: Virtual reality simulation training can improve technical skills during laparoscopic salpingectomy for ectopic pregnancy — https://pubmed.ncbi.nlm.nih.gov/17081183/
- See also: Assessment of technical skills transfer from the bench training model to the human model — https://pubmed.ncbi.nlm.nih.gov/10204564/
- See also: Description and validation of the Pelv-Sim: a training model designed to improve gynecologic minimally invasive suturing skills — https://pubmed.ncbi.nlm.nih.gov/18971133/